CLINICAL TRIAL: NCT00345501
Title: Iloprost for Prevention of Contrast-Mediated Nephropathy in High-Risk Patients With Preexisting Renal Dysfunction Undergoing a Coronary Procedure
Brief Title: Iloprost for Prevention of Contrast-Mediated Nephropathy in High-Risk Patients Undergoing Coronary Angiography and/or Intervention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Onassis Cardiac Surgery Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OCS IEC 265; EudraCT 2005-001887-30
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-08

CONDITIONS: Renal Insufficiency, Chronic; Coronary Angiography; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: contrast media; contrast nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Iloprost
  Interventions: Drug: Iloprost
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloprost — Iloprost 1ng/kg/min IV starting 1 hour before the procedure and continuing for 4 hours after its end
  Arms: 1
Drug: Placebo — Placebo IV (Normal saline) starting 1 hour before the procedure and continuing for 4 hours after its end
  Arms: 2

SUMMARY:
The prevention of contrast-mediated nephropathy (CMN), which accounts for considerable morbidity and mortality, remains a vexing problem. Contrast induced renal vasoconstriction is believed to play a pivotal role in the CMN mechanism. The aim of this study is to examine the efficacy of the prostacyclin analogue iloprost (dose 1ng/kg/min) in preventing CMN in high-risk patients undergoing a coronary procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically driven, non-emergent coronary angiography or intervention in our institution were eligible for inclusion if their serum creatinine concentration was ≥1.4 mg/dl (124 μmol/l) and/or their creatinine clearance was <60 ml/min on their most recent sample drawn within 1 month of the planned procedure

Exclusion Criteria:

* Circulatory shock for any reason, systolic blood pressure <95 mm Hg
* Known acute renal failure
* End-stage renal disease requiring dialysis
* Intravascular administration of a contrast medium within the previous 10 days
* Anticipated re-administration of contrast medium within the following 6 days
* Inability to administer intravenous hydration at least 4 h before the procedure or study medication at least 30 min before the procedure
* Primary intervention for acute infarction with ST elevation
* A procedure performed within 2 h of acute hospital admission

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2005-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
CMN is defined as an absolute increase of serum creatinine concentration of at least 0.5 mg/dl | 2-5 days after the procedure
or CMN is defined as a relative rise of at least 25% from baseline on the follow-up | blood sample drawn at 2-5 days after the procedure

SECONDARY OUTCOMES:
Differences in the progression of serum creatinine concentrations and creatinine clearance among the study groups | 2-5 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Spargias, MD, Principal Investigator — Onassis Cardiac Surgery Centre
Locations (1):
- Onassis Cardiac Surgery Centre, Athens, Greece

REFERENCES:
- [Derived] Spargias K, Adreanides E, Demerouti E, Gkouziouta A, Manginas A, Pavlides G, Voudris V, Cokkinos DV. Iloprost prevents contrast-induced nephropathy in patients with renal dysfunction undergoing coronary angiography or intervention. Circulation. 2009 Nov 3;120(18):1793-9. doi: 10.1161/CIRCULATIONAHA.109.863159. Epub 2009 Oct 19. PMID 19841299
- See also: Hospital Site — http://www.onasseio.gr